CLINICAL TRIAL: NCT04513314
Title: A Practical, Pilot, Randomized, Controlled Trial of Valproate Alone or in Combination With Quetiapine for Severe COVID-19 Pneumonia With Agitated Delirium
Brief Title: Valproate Alone or in Combination With Quetiapine for Severe COVID-19 Pneumonia With Agitated Delirium
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: coronavirus omicron variant infection typically not associated with delirium and agitation severely hampered recruitment.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Dominique Musselman, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20200851
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Hyperactive Delirium; Pneumonia, Viral
MeSH Terms: conditions — COVID-19; Pneumonia, Viral | interventions — Valproic Acid; Quetiapine Fumarate; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: study rater/outcomes assessor and participant will be ignorant of the treatment arm pharmacist and investigator will be aware of the treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Only Group (Active Comparator): Patients maintained with mechanical ventilation will be treated with standard of care after cessation of paralytic agents.
  Interventions: Other: Standard of Care
- Treatment Arm Group (Active Comparator): Patients maintained with mechanical ventilation will be treated with standard of care, plus Valproate on Days 1-7 after cessation of paralytic agents, and then augmented by the addition of Quetiapine beginning Days 3-7 if there are no improvement in RASS score.
  Interventions: Drug: Valproate; Drug: Quetiapine; Other: Standard of Care

INTERVENTIONS:
Drug: Valproate — Valproate sodium (enteral or intravenous) will be administered at a dosage of 10 to 15 mg/kg/day. The dosage may be increased by 5 to 10 mg/kg/week to achieve optimal clinical response. Ordinarily, optimal clinical response is achieved at daily doses below 60 mg/kg/day.
  Other Names: Depakote, Valproic acid
  Arms: Treatment Arm Group
Drug: Quetiapine — Enteral quetiapine dosing on Day 3: 25 mg to 50 mg twice daily. Increase in increments of 50 mg/day to 100 mg/day divided two on Days 4 and 5 to range of 50-400 mg/day by Day 7. Further adjustments can be made in increments of 25-50 mg twice a day, in intervals of not less than 2 days. Recommended dose range is 150-750 mg/day.
  Other Names: seroquel
  Arms: Treatment Arm Group
Other: Standard of Care — Standard of Care is a combination of IV dexmedetomidine (D), midazolam (M), ketamine (K) and propofol (P), at the discretion of treating physician.
  Other Names: Hospital Protocol

SUMMARY:
The primary purpose of this research is to determine whether Valproate alone, and in combination with Quetiapine, lowers confusion and agitation in persons with severe Corona Virus Disease (COVID)19 pneumonia during weaning from the breathing machine (ventilator). Though Valproate and Quetiapine are often given to persons with severe confusion with agitation, the purpose of this small research study is specifically for: a) persons infected with COVID 2019 on a ventilator whose agitation is not responding to the usual medications (like dexmedetomidine), and b) to reduce the time persons are treated with dexmedetomidine, which requires continuous close monitoring in an ICU.

DETAILED DESCRIPTION:
This is a pilot feasibility study involving a randomized, single-blind, controlled comparison scheme examining the efficacy and safety of standard of care (n=10) combined with valproate alone, and in combination with quetiapine (N=10) , in order to reduce the magnitude of agitation associated with COVID 19 delirium as assessed by the RASS scale when weaning from a ventilator, and reduce need for dexmedetomidine as assessed by number of doses of dexmedetomidine administered.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form by his or her legal/authorized representative
* Age ≥ 18 years at time of signing Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgement
* Hospitalized with COVID-19 pneumonia confirmed with World Health Organization (WHO) criteria (including an RNA test of any specimen, e.g. respiratory, blood, urine, stool, other bodily fluid) and evidence by chest X-ray or CT scan
* Fraction of inspired oxygen (Fi02) ≤ 0.40 and positive end-expiratory pressure (PEEP) ≤8 OR Fi02 ≤ 0.50 and PEEP ≤5
* Fi02 and PEEP ≤ values of previous day
* Patient has acceptable spontaneous breathing efforts (may decrease vent rate by 50% for 5 minutes to detect effort.)
* No neuromuscular blocking agents or blockade.
* RASS score initially at -3 ≤, rising to 3+ after initial attempt to wean from standard of care sedating medications
* Other investigational interventions may be permitted

Exclusion Criteria:

* Known severe allergic reactions to valproate or quetiapine
* History of hepatic encephalopathy or end-stage liver disease (Childs-Pugh class B or worse)
* Alcohol, or history of alcohol/substance dependence prior to admission
* Hx of dementia
* Treatment with an antipsychotic agent in the 30 days before ICU admission
* Baseline QT duration corrected (QTc) interval ≥ 500 msecs
* Pregnancy
* Suspected active bacterial, fungal, viral, or other infection (besides COVID-19)
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 X upper limit of normal (ULN) detected within 24 hours at screening or at baseline
* Absolute neutrophil count (ANC) < 1000/microliter (uL) at screening and baseline
* Platelet count < 50,000/uL at screening and baseline
* Individuals < 18 (infants, children, teenagers)
* Any serious medical condition or abnormality of clinical laboratory tests that, in the investigator's judgement, precludes the patient's safe participation in and completion of the study, e.g. active seizure disorder already receiving treatment with lamotrigine
* Informed consent could not be obtained from the legally authorized representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-28 (Estimated); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline RASS score of +3 or greater | Baseline, Day 7
  Richmond Agitation Sedation Scale (RASS) score ranges from +4 (combative) to 0 (alert & calm) to -5 (unarousable).

SECONDARY OUTCOMES:
Total dose of dexmedetomidine administered | Day 7
  Total dose of dexmedetomidine administered will be reported from baseline RASS score of +3 or greater.
Incidence of Treatment Emergent Adverse Events | Day 7
  Incidence of Treatment Emergent Adverse Events will include:
  * QTc duration > 470 msecs.
  * Increase in Liver Function Tests to a Grade 3 or higher using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
  * Suicidality reported as having a score of moderate or high risk using the Columbia-Suicide Severity Rating Scale Screening (C-SSRS). C-SSRS is a calculated risk assessment tool that scores suicidality from no risk to high risk.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique L Musselman, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goel D, Srivastava A, Aledo-Serrano A, Krishnan A, Vohora D. Pharmacotherapy for SARS-CoV-2 and Seizures for Drug Repurposing Presumed on Mechanistic Targets. Curr Mol Pharmacol. 2022;15(6):832-845. doi: 10.2174/1874467214666211013122528. PMID 34645381